CLINICAL TRIAL: NCT02621099
Title: First Use of a Hybrid Gamma Camera for Sentinel Lymph Node Localisation in Patients Undergoing Surgery for Primary Breast Cancer
Brief Title: Hybrid Gamma Camera in Breast Surgery
Acronym: HICAM
Status: Withdrawn | Type: Observational
Why Stopped: The study was withdrawn due to the CE mark of the device was not yet granted during the specified period.
Sponsor: University of Nottingham (Other)
Collaborators: Innovate UK (Other Government)
Responsible Party: Sponsor
Other Study IDs: 15096
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer
Keywords: handheld gamma camera
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Hybrid optical-gamma imaging — Acquisition of images using the camera as additional steps to the standard SLNB procedures.

SUMMARY:
A novel hand held hybrid optical-gamma camera (hereinafter referred to as the "camera") has been developed and can be used to image radiotracer distribution at the patient bedside. This study aims to evaluate the imaging capabilities of the camera in patients attending surgery for sentinel lymph node biopsy (SLNB) procedure. It is anticipated that this could improve the accuracy and simplify sentinel lymph node detection by providing fused optical and gamma imaging.

DETAILED DESCRIPTION:
This is a single centre prospective, non-randomised and non-blinded research project using the camera in the operating theatre in addition to the standard gamma surgical probe for assessing lymph node involvement in breast cancer patients undergoing surgery for their disease. The duration of the study is 1 year.

The purpose of the trial will be to determine if the camera can be used for the localisation of sentinel lymph nodes during the SLNB procedure and to compare detection rates of sentinel lymph node(s) with the standard method using the gamma probe.

Study Plan:

This study will not alter the standard SLNB procedures provided by the healthcare provider. The camera will be used to acquire images in the axillary and parasternal regions as additional steps to the standard SLNB procedures. No invasive actions are performed. Images obtained using the camera in this study will include gamma, optical and fused gamma/optical images in each acquisition. In additional to the intraoperative imaging study using the camera system, a subjective assessment by questionnaire will be carried out amongst the surgeons to obtain their feedback.

Statistics:

For the quantitative analysis, the distribution of continuous variables will be summarised using mean and standard deviation (if normally distributed) or median and range (if not normally distributed); distribution of categorical variables will be summarised by presenting the number and percentages that falling into each categories. Missing data will be recorded. SPSS will be used to manage the data. The detection rate of both detection methods (camera versus standard techniques) will be tabulated as binary data (yes/no). Validity analysis will be computed for sensitivity, specificity, positive predictive value and negative predictive value. Also Kappa (categorical data) method will be used to examine the agreement between two methods. Good agreement will be claimed if the value of kappa between 0.81 and 1.00.

Sample size:

The calculated sample size is 53 participants. It has been calculated using nQuery Advisor® 6.0 with the goal to make conclusion using agreement. The sample size has the 80% power to pick up ҡ1 = 0.410 or greater.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age > 18 years
* Scheduled for a Sentinel Lymph Node Biopsy procedure for breast cancer
* Has capacity to provide written 'informed consent'

Exclusion Criteria:

Non-English speaking patients who have had:

* a nuclear medicine procedure with administration of a radiopharmaceutical within 72 hours prior to the procedure;
* prior systemic therapy for the breast cancer being scheduled for sentinel node biopsy (e.g. neoadjuvant chemotherapy and primary endocrine therapy).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients scheduled for a sentinel lymph node biopsy (SLNB) procedure for breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2017-02 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Agreement of detection rate between the camera and standard gamma probe in the SLNB | 12 months

SECONDARY OUTCOMES:
Symmetry of detection rate between the camera and gamma probe in the SLNB | 12 months
Additional information obtained by the camera in the SLNB | 12 months
Additional information on internal mammary node detection | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kwok Leung Cheung, Study Chair — University of Nottingham
Locations (1):
- Royal Derby Hospital, Derby, United Kingdom

REFERENCES:
- [Background] Ng AH, Clay D, Blackshaw PE, Bugby SL, Morgan PS, Lees JE, Perkins AC. Assessment of the performance of small field of view gamma cameras for sentinel node imaging. Nucl Med Commun. 2015 Nov;36(11):1134-42. doi: 10.1097/MNM.0000000000000377. PMID 26352214
- [Background] Bugby SL, Lees JE, Bhatia BS, Perkins AC. Characterisation of a high resolution small field of view portable gamma camera. Phys Med. 2014 May;30(3):331-9. doi: 10.1016/j.ejmp.2013.10.004. Epub 2013 Nov 10. PMID 24225012
- [Background] Bhatia BS, Bugby SL, Lees JE, Perkins AC. A scheme for assessing the performance characteristics of small field-of-view gamma cameras. Phys Med. 2015 Feb;31(1):98-103. doi: 10.1016/j.ejmp.2014.08.004. Epub 2014 Nov 13. PMID 25440940
- [Background] Lees, J.E., et al., A small field of view camera for hybrid gamma and optical imaging. Journal of Instrumentation, 2014. 9: p. C12020.
- [Background] Lees, J.E., et al., A high resolution Small Field Of View (SFOV) gamma camera: a columnar scintillator coated CCD imager for medical applications. Journal of Instrumentation, 2011. 6.